CLINICAL TRIAL: NCT05718362
Title: Investigation of the Effect of Ayres Sensory Integration Therapy on Occupational Performance in Children With Autism Spectrum Disorder: A Randomized Control
Brief Title: Ayres Sensory Integration Therapy on Occupational Performance in Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Zeynep Çorakcı Yazıcıoğlu, Lecturer, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CORAKCİ-001
Record Dates: First submitted 2023-01-06; First posted 2023-02-08 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Autism Spectrum Disorder
Keywords: Ayres Sensory Integration; Occupational Performance
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: 2 groups will be formed as study and control. A simple random distribution will be made when creating groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Ayres Sensory Integration Therapy and Home Program
  Interventions: Behavioral: Ayres Sensory Integration Therapy; Behavioral: Home Program
- Control Group (Active Comparator): Home Program
  Interventions: Behavioral: Home Program

INTERVENTIONS:
Behavioral: Ayres Sensory Integration Therapy — It is an intervention method whose effectiveness is questioned. It is a therapy program applied according to Ayres Sensory Integration Fidelity Measure.
  Arms: Intervention Group
Behavioral: Home Program — These are the activities created for the participants (both intervention and control groups) and to be done in the home environment.

SUMMARY:
Ayres Sensory Integration (ASI) Therapy is an individualized intervention designed to address specific underlying sensorimotor issues that may affect children's performance during daily routines and occupations. The intervention takes place in the context of play, emphasizes the active participation of the child, involves a collaborative relationship between the occupational therapist and the child, and focuses on participation-oriented outcomes that are collected at regular intervals throughout the intervention program. In general, its content is to improve the child's occupational performance.

The program, which will be carried out in accordance with the Ayres Sensory Integration Fidelity Measure®, it is aimed to reduce the autism-specific symptoms of the child with autism and the dependence of the child on the caregiver in self-care activities. It is predicted that this whole process will increase the participation and his performance of the child with autism in his occupations related to his daily life.

H0: Ayres Sensory Integration Therapy has no effect on the occupational performance of the child with autism spectrum disorder.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with Autism Spectrum Disorder according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition
* Level 1 (requiring support) and Level 2 (requiring substantial support) are severity levels for Autism Spectrum Disorder
* Age at first and second test between 3 years and 10 years

Exclusion Criteria:

* Accompanying neurodevelopmental, psychiatric, neurological or physical diagnosis

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2023-01-06 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Occupational Performance | 4 months
  Occupational performance will be evaluated with Canadian Occupational Performance Measure (COPM). The measure is a goal-oriented, individualized, client-centered tool in which participants can set different goals in self-care, productivity, and leisure.
  * The measure is a semi-structured assessment applied to determine the daily activities that participants have difficulty with.
  * All activities said by the participants are scored between 1-10 points and the first five activities are selected.
  * These activities are also scored between 1-10 points according to performance and satisfaction.
  * Scores are compared by applying the same scale after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Çorakcı, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakıf University, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Corakci Yazicioglu Z, Bumin G. Occupational Therapy Using Sensory Integration for Enhancing Occupational Performance in Children with Autism: A Randomized Controlled Trial. J Autism Dev Disord. 2025 Jul 25. doi: 10.1007/s10803-025-06970-1. Online ahead of print. PMID 40711707